CLINICAL TRIAL: NCT03950219
Title: CUlturally Sensitive TOols and Methods for Ethnic Minorities (CUSTOM): Building Bridges Between Theory and Practice in Diabetes Self-management Education and Support
Brief Title: CUlturally Sensitive TOols for Ethnic Minorities in Diabetes Self-management Education and Support
Acronym: CUSTOM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Center for Diabetes, Copenhagen Municipality (Other Government)
Responsible Party: Principal Investigator, Nana Folmann Hempler, Team leader and senior researcher, Steno Diabetes Center Copenhagen
Other Study IDs: CUSTOM
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes self-management; Diabetes Education; Ethnic minorities; Patient empowerment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention, Centre for Diabetes or local setting: Group-based course in diabetes education including 6 sessions of approximately 3 hours. Sessions are constructed around themes such as; diabetes knowledge and complication, mental health, diet, physical activity, Ramadan, medicine and include practical exercises such as blood sugar measurements, walking etc.
- Usual care: Usual care in 5 municipalities in the west area of Copenhagen
  Interventions: Other: Group course

INTERVENTIONS:
Other: Group course — Education and support
  Groups: Usual care

SUMMARY:
The CUSTOM research project represents a complex intervention. The project aim of the intervention is, through the delivery of culturally sensitive Diabetes self-management education and support, to support ethnic minorities with type 2 diabetes in making health-promoting decisions about their care and gaining insight into their goals, values and motivation to improve their daily diabetes self-management. The target group comprises ethnic minorities whose native language is Arabic, Urdu or Turkish.

DETAILED DESCRIPTION:
The CUSTOM research project represents a complex intervention. The project aim of the intervention is, through the delivery of culturally sensitive DSMES, to support ethnic minorities with type 2 diabetes in making health-promoting decisions about their care and gaining insight into their goals, values and motivation to improve their daily diabetes self-management. The target group comprises ethnic minorities whose native language is Arabic, Urdu or Turkish. The intervention has been developed in collaboration with the target group and health care professionals from Centre for Diabetes (CfD) in Copenhagen Municipality.

CUSTOM will explore feasibility and effectiveness of the intervention including the mechanisms through which outcomes occur and contexts where outcomes are likely to be replicable. The intervention builds on the framework of complex interventions(26), and is designed as an pragmatic randomised controlled trial in three arms.

Focus on fidelity, appropriateness and acceptability of the developed intervention.

* What factors and structures are necessary to facilitate DSMES access and retention among the target group?
* Which methods and tools supporting diabetes decision making and problem solving are acceptable and feasible among the target group?
* What educational strategies promote Health Care Professionals' (HCPs') communication with the target group?

Focus on exploring effectiveness of the intervention, the mechanisms through which outcomes occur and contexts where outcomes are likely to be replicable.

* To what extent does the intervention lead to better outcomes (e.g., HbA1c and participant-reported outcomes) than 'usual care' for the target group and what mechanisms for the effect of the intervention can be identified? And are there differences according to the setting, of which the intervention is delivered; a) in a community health centre and b) a local community setting.
* What characterizes contexts that are most conducive to positive outcomes?
* What barriers and possibilities exist related to implementing culturally sensitive DSMES in different municipal settings targeting ethnic minority groups?
* Which contextual factors determine whether the identified mechanisms lead to intended outcomes?
* What are the long-term effects of the intervention on measured outcomes?

Study design CUSTOM is considered a complex intervention due to many interacting components in its design, complex behaviour changes in those delivering and receiving the intervention, many stakeholders, and highly variable outcomes. The trial will be undertaken as a pragmatic trial using cluster randomisation.

The trial will be tested in three arms: Participants will be randomised into 3 arms Group A: Centre for Diabetes, Copenhagen Municipality, n = 103 Group B: Local community setting in Tingbjerg, Copenhagen Municipality, n = 103 Group C: Usual care in the west area of Copenhagen, municipalities of Høje-Taastrup, Hvidovre, Albertslund, Brøndby and Ishøj, n = 103 Figure 1 Study Design 9. Interventions 9.1 Group A and B: Group A and B will receive the same interventions but in different contexts - a local community setting and a diabetes care centre. The intervention will be pilot tested in the local community and if necessary adjusted to local contexts.

Using a design-based research, the intervention has been developed in collaboration with researchers, the target group and healthcare professionals from Centre for Diabetes (CfD) in Copenhagen Municipality.

The group-based course will include 6 sessions of approximately 3 hours. Sessions are constructed around themes such as; diabetes knowledge and complication, mental health, diet, physical activity, Ramadan, medicine and include practical exercises such as blood sugar measurements, walking etc. The healthcare professionals delivering the education consists of an interdisciplinary team of both a nurse, dietitian, physiotherapist, a translator and a peer educator.

The CUSTOM intervention consists of three elements: philosophy/values, educator behaviours and 12 specific dialogue tools. These three elements are all equally important in the organisation and completion of a good and culturally sensitive diabetes education targeting ethnic minorities. The intervention is based on the concept CUSTOM which is developed with regards to the healthcare professionals' approaches, methods and existing educational activities. The concept consists of 12 health education tools accompanied by a comprehensive guide. The success of the tools developed in CUSTOM rely on the values held by the suppliers of the education and by the health care professional's competences to apply the specific dialogue tools.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes
* Ability to give written consent
* Ability and willingness to attend and participate in a group-based education programme.
* First language is Arabic, Turkish or Urdu.

Exclusion Criteria:

* Physical illness that could seriously reduce their life expectancy and ability to participate in the trial
* Mental illness that could reduce their ability to participate in the trial
* Significant alcohol or substance misuse which could limit the participants ability to participate in the trial
* A primary diagnosis of learning disability
* Pregnancy, breastfeeding or plans of pregnancy during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Referred to rehabilitation by the GP and has type 2 diabetes
Sampling Method: Probability Sample
Enrollment: 309 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Well-being | 6 months
  questionnaire
diabetes self-management | 6 months
  questionnaire
HbA1c | 6 months
  blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Nana F Hempler, PhD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Centre for Diabetes, Copenhagen, Denmark